CLINICAL TRIAL: NCT01943487
Title: A Phase 1, Open-label, One-sequence Study to Assess the Effect of Verapamil on the Steady State Pharmacokinetics of Solifenacin and Tamsulosin Administered as a Combination Tablet EC905 in Healthy Male Subjects.
Brief Title: A Study to Evaluate Whether Verapamil Has an Effect on the Uptake and Elimination of Solifenacin and Tamsulosin When Administered in a Combination Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 905-CL-078; 2009-010841-29 (EudraCT Number)
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Drug-Drug Interaction (DDI); Healthy Subjects
Keywords: Phase I; Verapamil; Tamsulosin OCAS; Solifenacin; Pharmacokinetics; EC905
MeSH Terms: interventions — Solifenacin Succinate; Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1: verapamil + EC905 (Experimental)
  Interventions: Drug: EC905; Drug: verapamil

INTERVENTIONS:
Drug: EC905 — Oral
  Other Names: tamsulosin OCAS and solifenacin
Drug: verapamil — Oral

SUMMARY:
This study investigates the effect of the co-administration of verapamil on the steady-state pharmacokinetics (PK) of solifenacin succinate and tamsulosin given as a combination tablet, EC905.

DETAILED DESCRIPTION:
The effect of the co-administration of verapamil on the steady state PK of solifenacin succinate and tamsulosin HCl OCAS (Oral Controlled Absorption System) is evaluated in this study.

Verapamil has been chosen to represent the effect of moderate CYP3A4 inhibitors on the combined administration of solifenacin and tamsulosin given as combination tablet EC905.

Subjects are admitted to the clinic on Day -1. From Days 1-10, they receive one daily dose of EC905 to obtain steady state, followed by 20 days (Days 11-30) combined dosing of EC905 and verapamil.

On Day 10 a 24-hour PK profile is obtained for solifenacin/tamsulosin. After the last dosing on Day 30, a post-dose 24-hour PK profile for solifenacin/tamsulosin and verapamil is obtained.

Additionally, vital signs, safety ECG (Electrocardiogram) measurements, safety laboratory assessments, adverse events and concomitant medications are monitored throughout the investigational period.

Subjects return for an ESV (End of Study Visit) 10 days after the last dosing.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 18.5 and 30.0 kg/m2, inclusive

Exclusion Criteria:

* Known or suspected hypersensitivity to EC905 or any of the components of the formulation used
* Known or suspected hypersensitivity to verapamil or any of the components of the formulation used
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampin) in the 3 months prior to admission to the Clinical Unit

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of tamsulosin OCAS in plasma: AUCtau | Predose, Days 1, and 7-10
  AUCtau (area under the plasma concentration-time curve during the time interval between consecutive dosing)
Pharmacokinetics of solifenacin in plasma: AUCtau | Predose, Days 1, and 7-10
  AUCtau (area under the plasma concentration-time curve during the time interval between consecutive dosing)
Pharmacokinetics of tamsulosin OCAS in plasma: Cmax | Predose, Days 1, and 7-10
  Cmax (maximum concentration)
Pharmacokinetics of solifenacin in plasma: Cmax | Predose, Days 1, and 7-10
  Cmax (maximum concentration)

SECONDARY OUTCOMES:
Pharmacokinetics of combined doses of tamsulosin OCAS and solifenacin in steady state, and verapamil | Predose, Days 27-30
  Plasma: Ctrough (trough concentration), tmax (time to attain Cmax), CL/F (apparent total body clearance), PTR (peak trough ratio) Urine: AUCtau, Cmax, Ctrough, CL/F, tmax
Safety and tolerability of the interaction between combined doses of tamsulosin OCAS and solifenacin, and verapamil | Screening to ESV (10 days after the last dosing)
  AE (adverse events), clinical laboratory tests, vital signs, ECG, physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- SGS Aster, Paris, France